CLINICAL TRIAL: NCT04436393
Title: Guardant360® Related Clinical Outcomes in Patients Who Share Medical Records-Breast Cancer
Acronym: GRECO-B
Status: Completed | Type: Observational
Sponsor: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-BR-003
Record Dates: First submitted 2020-04-16; First posted 2020-06-18 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Breast Cancer: Patients with diagnosis of advanced breast cancer
  Interventions: Diagnostic Test: Guardant360 test

INTERVENTIONS:
Diagnostic Test: Guardant360 test — tumor cfDNA testing

SUMMARY:
The purpose of this study is to observe the routine clinical care of patients who have been diagnosed with breast cancer and have undergone Guardant360 testing.

DETAILED DESCRIPTION:
Patients who have been diagnosed with breast cancer and have undergone Guardant360 testing will be approached regarding participation in the study. After being informed about the study and potential risks, all patients providing informed consent and access to their medical records, will provide a list of their health care providers related to their cancer treatment. Data related to their routine clinical care will be abstracted from medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years of age and older) with a diagnosis of breast cancer
2. Guardant360 test results released to the patient's physician no less than 14 days prior to initial patient contact
3. Patient has previously provided contact information (either email or phone) to Guardant Health
4. Able and willing to complete the electronic informed consent process
5. Must have access to a computer terminal or personal computing device
6. Willingness to consent to the release of medical records

Exclusion Criteria:

1. Unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects located in the United States that have undergone Guardant360 testing as part of their routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 18 months post Guardant360 testing
  The Primary Outcome measure is a composite endpoint of: overall survival, progression events, and subjects lost-to-follow-up
  Overall Survival is the length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Progression Events | 18 months post Guardant360 testing
  The Primary Outcome measure is a composite endpoint of: overall survival, progression events, and subjects lost-to-follow-up
  Progression events (or progression-free survival) is the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Subject Lost-to-Follow-Up | 18 months post Guardant360 testing
  The Primary Outcome measure is a composite endpoint of: overall survival, progression events, and subjects lost-to-follow-up
  The length of time from date of study consent to date subject exited study prematurely due being considered lost-to-follow-up (ex. lack of response following consent)

SECONDARY OUTCOMES:
Rate of biomarker discovery | 18 months post Guardant360 testing
  Assess the rate of biomarker discovery compared to tumor genotyping results
Time to Next Treatment | 18 months post Guardant360 testing
  Assess time to next treatment decision compared to tumor genotyping results
Real-world Time to Tumor Progression | 18 months post Guardant360 testing
  Documented tumor progression either clinically or radiologically
Real-world Overall Survival | 18 months post Guardant360 testing
  Date of death per clinical record or secondary sources (e.g. national death registries)
Demographics | 18 months post Guardant360 testing
  Descriptive statistics of patient demographics

CONTACTS AND LOCATIONS:
Overall Officials: Victoria M Raymond, M.S., Principal Investigator — Guardant Health, Inc.
Locations (1):
- Guardant Health, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No